CLINICAL TRIAL: NCT06008860
Title: A Pilot Clinical Evaluation of Astepro® Nasal Spray for Management of Early SARS-CoV-2 Infection
Acronym: COVID-19
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB22-1144
Record Dates: First submitted 2023-08-21; First posted 2023-08-24 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — azelastine

STUDY DESIGN:
Intervention Model Description: All subjects will be sent an instructional video and be given written instructions which will educate them on how to use the drug or placebo nasal spray. Patients will follow the dosing instructions for Astepro® 0.15% nasal spray.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind clinical trial. Randomization schedules will be generated and stratified by age (18-30, 31--40, 41-50, and ≥50 years) and sex, using computer-generated random numbers and alternating block sizes. Only the study statistician will have access to the randomization lists. The assigned treatment for each study subject will be obtained via REDCap. The Investigational Drug Service (IDS) pharmacy will be used to distribute the drug or placebo as provided by Bayer. The pharmacy will also help to coordinate and track randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Primary Cohort - Azelastine (Other): This is a double-blind clinical trial. All subjects will be sent an instructional video and be given written instructions which will educate them on how to use the drug or placebo nasal spray. Patients will follow the dosing instructions for Astepro® 0.15% nasal spray.
  Interventions: Drug: Experimental: Primary Cohort
- Primary Cohort - Placebo (Placebo Comparator): This is a double-blind clinical trial. A Placebo will be provided by Bayer which features similar color and packaging. Both groups will also undergo recommendations for supportive care, which will be standardized. Any patients who develop severe disease will be given instructions for escalation of care.
  Interventions: Other: Placebo Comparator: Primary Cohort - Placebo

INTERVENTIONS:
Drug: Experimental: Primary Cohort — Astepro (azelastine) is a second generation antihistamine, as well as an anti-inflammatory and mast cell stabilizer8. It is available as a 0.1% and 0.15% nasal spray by prescription in the USA and over-the-counter in the European Union (EU). Dosing for adults and adolescents 12 years and older is 1 or 2 sprays per nostril twice daily (0.1%) or 2 sprays per nostril once daily (0.15%)9. It is approved by the FDA for treatment of seasonal allergic rhinitis symptoms (rhinorrhea, sneezing, and nasal pruritus) in adults and children 2 years and older, perennial allergic rhinitis in adults and children ages 6 months and older, and the symptoms of vasomotor rhinitis (rhinorrhea, nasal congestion and postnasal drip) in adults and adolescents 12 years and older9.
  Other Names: azelastine
  Arms: Primary Cohort - Azelastine
Other: Placebo Comparator: Primary Cohort - Placebo — A Placebo will be provided by Bayer which features similar color and packaging as azelastine.
  Arms: Primary Cohort - Placebo

SUMMARY:
The study team proposes to evaluate the efficacy of Astepro® 0.15% nasal spray in treating SARS-CoV-2 infection in adults through a pilot and feasibility clinical trial at the University of Chicago.

DETAILED DESCRIPTION:
In this study, the study team aims to re-confirm the utility of this medication for use in Covid-19 to decrease the significant impact on quality of life, symptoms, infectivity, and occupation. plan to recruit vaccinated adults immediately upon Covid-19 diagnosis at one major Chicago University and follow viral load as a primary outcome in those randomized to receive Astepro® vs. placebo. Subjects who have a home antigen test or polymerase chain reaction (PCR) positive diagnosis of Covid-19 will be enrolled in the study. Viral load will be assessed at Day -1, day of presentation, followed by self-collected saliva over the subsequent 10 days in patients getting either azelastine or placebo.

Specific Aims

To address this hypothesis, the study team is investigating the following specific aims:

1. Compare the trajectories of SARS-CoV-2 viral load in the upper airway of adults with new onset Covid-19 randomized to receive azelastine at standard rhinitis dosing (n=70) or placebo (n=70) over 10 days. The study team will target early disease (immediately upon diagnosis), mild severity in outpatients (facilitating study participation and self-sample collection), and pragmatic, receptive target populations (volunteers living nearby).
2. Determine if there is a decrease in R0 in Covid-19 positive patients and their closest contacts The study team hypothesizes that less new covid infections will be observed among close contacts who co-habitate with subjects randomized to the Astepro (azelastine) arm.
3. Determine whether treatment with azelastine improves pertinent clinical parameters in these subjects. Rates, durations, and intensities of key symptoms will be captured using existing, low burden data collection instruments that meet FDA guidelines. All sample and data collection, including validated, objective olfactory testing, will be contactless, minimizing risk.
4. Assess and quantitate side effects, subject satisfaction, and tolerability of azelastine in this setting. Given the heterogeneous nature of Covid-19, the study team will assess the feasibility of this treatment from the patient standpoint, including qualitative and quantitative feedback, to inform future trials and scaling.

ELIGIBILITY:
Inclusion Criteria (Primary Cohort):

* 18 and up
* Ability to consent
* Have a Covid-19 positive saliva sample prior to the start of treatment; or positive rapid antigen test at home confirmed via first COVID-19 positive saliva sample
* Ability to follow the study instructions and adhere to the study procedures
* Ability to provide every other day saliva samples throughout the study period 10 days, and report symptoms
* Subjects that have been vaccinated for Covid-19
* Does not have any symptoms or only experiencing mild symptoms of Covid-19 (e.g., such as fever below a threshold or no fever, or without severe cough, among others).

Inclusion Criteria (Close Contacts):

* Ability to consent
* Ability to follow the study instructions and report side effects
* Ability to provide saliva samples throughout the study period
* Subjects that have been vaccinated for Covid-19.

Exclusion Criteria (Primary Cohort):

* Women who are breastfeeding, pregnant, or who plan to become pregnant
* Contradictions to intranasal azelastine (known hypersensitivity)
* Use of other Covid-19 treatments (steroids, convalescent plasma, therapeutic antibodies, etc.)
* Intranasal, corticosteroid, immunomodulator, or other medication use which can change the effect of Astepro.
* Prior Covid infection greater than 5 and less than 30 days before enrollment
* Subjects who have been involved with any other research study within the last 30 days.
* A prior hypersensitivity to olopatadine (Patanase), diphenhydramine, hydroxyzine.

Subjects that have not been vaccinated for Covid-19. Subjects that have moderate to severe COVID-19 symptoms, or signs of meeting indications (e.g.

Shortness of Breath, chest pains) for urgent or emergent therapy (these subjects will be advised to seek emergency medical assistance).

Exclusion Criteria (Close Contacts)

* Prior Covid infection less than 30 days or greater 5 days prior to enrollment in study
* Use of other Covid-19 treatments
* Having a positive rapid home or PCR COVID test prior to the positive test for the primary cohort subject they're associated with
* Involved with any other research study within the last 30 days
* Subjects that have not been vaccinated for Covid-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Astepro for use in managing Covid-19 symptoms and assessing viral load in participants.. | Baseline (Day -1) through Day 10
  The primary cohort will be followed while utilizing study drug or placebo to evaluate the outcomes and saliva collection to follow viral load.

SECONDARY OUTCOMES:
Rate of Covid-19 infectivity in primary cohorts close contacts | Day 1, Day 11
  Saliva will be collected from close contacts to assess any changes in Covid-19 infectivity.
Change from baseline in upper respiratory symptoms and Quality of Life, as measured by the WURSS44 survey | Primary Cohort: Baseline (Day -1) through Day 10, Close Contact Cohort: Day 1 and Day 11
  WURSS44 is illness-specific quality of life instrument, designed to assess the negative impact of viral acute upper respiratory infection.
Change from baseline symptoms and quality of life utilizing the All of Us Research Program Covid-19 Participant Experience (COPE) survey | Primary Cohort: Baseline (Day -1) through Day 10, Close Contact Cohort: Day 1 and Day 11
  All of Us Research Program Covid-19 Participant Experience (COPE) survey is utilized to assess the health impact of Covid-19.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Baird, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wiersinga WJ, Rhodes A, Cheng AC, Peacock SJ, Prescott HC. Pathophysiology, Transmission, Diagnosis, and Treatment of Coronavirus Disease 2019 (COVID-19): A Review. JAMA. 2020 Aug 25;324(8):782-793. doi: 10.1001/jama.2020.12839. PMID 32648899
- [Background] Johns Hopkins University & Medicine. Coronavirus Resource Center. https://coronavirus.jhu.edu/. Accessed 01/26/2021.
- [Background] Palacios R, Patino EG, de Oliveira Piorelli R, Conde MTRP, Batista AP, Zeng G, Xin Q, Kallas EG, Flores J, Ockenhouse CF, Gast C. Double-Blind, Randomized, Placebo-Controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of treating Healthcare Professionals with the Adsorbed COVID-19 (Inactivated) Vaccine Manufactured by Sinovac - PROFISCOV: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Oct 15;21(1):853. doi: 10.1186/s13063-020-04775-4. PMID 33059771
- [Background] Rogosnitzky M, Berkowitz E, Jadad AR. Delivering Benefits at Speed Through Real-World Repurposing of Off-Patent Drugs: The COVID-19 Pandemic as a Case in Point. JMIR Public Health Surveill. 2020 May 13;6(2):e19199. doi: 10.2196/19199. PMID 32374264
- [Background] Beigel JH, Tomashek KM, Dodd LE, Mehta AK, Zingman BS, Kalil AC, Hohmann E, Chu HY, Luetkemeyer A, Kline S, Lopez de Castilla D, Finberg RW, Dierberg K, Tapson V, Hsieh L, Patterson TF, Paredes R, Sweeney DA, Short WR, Touloumi G, Lye DC, Ohmagari N, Oh MD, Ruiz-Palacios GM, Benfield T, Fatkenheuer G, Kortepeter MG, Atmar RL, Creech CB, Lundgren J, Babiker AG, Pett S, Neaton JD, Burgess TH, Bonnett T, Green M, Makowski M, Osinusi A, Nayak S, Lane HC; ACTT-1 Study Group Members. Remdesivir for the Treatment of Covid-19 - Final Report. N Engl J Med. 2020 Nov 5;383(19):1813-1826. doi: 10.1056/NEJMoa2007764. Epub 2020 Oct 8. PMID 32445440
- [Background] World Health Organization. An international randomised trial of additional treatments for COVID-19 in hospitalised patients who are all receiving the local standard of care. https://www.who.int/publications/m/item/an-international-randomised-trial-of-additional-treatments-for-covid-19-in-hospitalised-patients-who-are-all-receiving-the-local-standard-of-care.
- [Background] Bernstein JA. Azelastine hydrochloride: a review of pharmacology, pharmacokinetics, clinical efficacy and tolerability. Curr Med Res Opin. 2007 Oct;23(10):2441-52. doi: 10.1185/030079907X226302. PMID 17723160
- [Background] U.S. Food & Drug Administration. Astelin Nasal Spray Full Prescribing Information. https://www.accessdata.fda.gov/drugsatfda_docs/label/2015/022203s010s011lbl.pdf. Accessed 01/26/2021.
- [Background] Reznikov LR, Norris MH, Vashisht R, Bluhm AP, Li D, Liao YJ, Brown A, Butte AJ, Ostrov DA. Identification of antiviral antihistamines for COVID-19 repurposing. Biochem Biophys Res Commun. 2021 Jan 29;538:173-179. doi: 10.1016/j.bbrc.2020.11.095. Epub 2020 Dec 3. PMID 33309272
- [Background] Freedberg DE, Conigliaro J, Wang TC, Tracey KJ, Callahan MV, Abrams JA; Famotidine Research Group. Famotidine Use Is Associated With Improved Clinical Outcomes in Hospitalized COVID-19 Patients: A Propensity Score Matched Retrospective Cohort Study. Gastroenterology. 2020 Sep;159(3):1129-1131.e3. doi: 10.1053/j.gastro.2020.05.053. Epub 2020 May 22. No abstract available. PMID 32446698
- [Background] Ghosh R, Chatterjee S, Dubey S, Lavie CJ. Famotidine Against SARS-CoV2: A Hope or Hype? Mayo Clin Proc. 2020 Aug;95(8):1797-1799. doi: 10.1016/j.mayocp.2020.05.027. Epub 2020 Jun 6. No abstract available. PMID 32753153
- [Background] Ennis M, Tiligada K. Histamine receptors and COVID-19. Inflamm Res. 2021 Jan;70(1):67-75. doi: 10.1007/s00011-020-01422-1. Epub 2020 Nov 18. PMID 33206207
- [Background] Laird NM, Ware JH. Random-effects models for longitudinal data. Biometrics. 1982 Dec;38(4):963-74. PMID 7168798
- [Background] To KK, Tsang OT, Leung WS, Tam AR, Wu TC, Lung DC, Yip CC, Cai JP, Chan JM, Chik TS, Lau DP, Choi CY, Chen LL, Chan WM, Chan KH, Ip JD, Ng AC, Poon RW, Luo CT, Cheng VC, Chan JF, Hung IF, Chen Z, Chen H, Yuen KY. Temporal profiles of viral load in posterior oropharyngeal saliva samples and serum antibody responses during infection by SARS-CoV-2: an observational cohort study. Lancet Infect Dis. 2020 May;20(5):565-574. doi: 10.1016/S1473-3099(20)30196-1. Epub 2020 Mar 23. PMID 32213337
- [Background] Hedeker D. Multilevel Models for Ordinal and Nominal Variables. In: Leeuw Jd, Meijer E, eds. Handbook of Multilevel Analysis. New York, NY: Springer New York; 2008:237-274.